CLINICAL TRIAL: NCT02853201
Title: Monitoring Intercostal Muscles After Extubation
Acronym: MIME
Status: Completed | Type: Observational
Sponsor: Unity Health Toronto (Other)
Responsible Party: Principal Investigator, Laurent Brochard, Clinician Scientist, Unity Health Toronto
Other Study IDs: REB# 16-161
Record Dates: First submitted 2016-07-29; First posted 2016-08-02 (Estimated); Last update posted 2018-04-10 (Actual); Status verified 2018-04

CONDITIONS: Respiratory Insufficiency
Keywords: Extubation; Intercostal Muscles; Diaphragm; Sternocleidomastoid Muscle
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Mechanical ventilation is a life-saving treatment for critically ill patients who are unable to breathe on their own. At the time of recovery, separation from the ventilator is performed without difficulty for the majority of patients. However, approximately 15% of patients experience extubation failure, i.e. they are re-intubated after extubation within a period of 48 hours to 7 days. Patients who fail extubation are exposed to a longer duration of mechanical ventilation, higher rates of ventilator-acquired pneumonia, higher morbidity, and higher ICU mortality. Therefore, it is of relevant importance for clinicians to identify patients who are at risk of extubation failure as soon as ventilation has been discontinued. However, current clinical assessment has poor predictive performance: some physiological variables can be helpful but can only be obtained invasively using esophageal and gastric catheters.

Using ultrasound measurements to assess the activity of the respiratory muscles could be of particular interest for this purpose. By showing an early recruitment of the accessory muscles as well as diaphragm dysfunction or hyperactivity, ultrasounds could help clinicians pay greater attention to such patients and therefore try to apply specific therapeutics. There are several advantages to ultrasounds: they are non-invasive, available in most intensive care units, and previous studies have reported reasonable reliability of the measurements.

In the present study, we aim to assess the contractility of the respiratory muscles (diaphragm, intercostal, and sternocleidomastoid) using ultrasounds to identify patients who may be at risk of extubation failure and/or ICU readmission.

DETAILED DESCRIPTION:
This study is a single centre, prospective, physiologic study in extubated patients (n = 110) to assess the contractility of the diaphragm, intercostal, and sternocleidomastoid muscles. The purpose is to determine whether employing ultrasounds early after extubation is a useful diagnostic tool to identify patients who may be at risk of extubation failure and/or intensive care unit (ICU) re-admission. The study will be performed in the Medical-Surgical ICU of St. Michael's Hospital.

Once the clinical team has decided to extubate the patient, the research team will approach the patient for consent (if capable) or the patient's substitute decision maker. Demographic information will be extracted from the medical chart and entered into the study case report form (CRF). Ultrasounds of the diaphragm, intercostal, and sternocleidomastoid muscles will be performed within 2 hours of extubation and repeated within 24 hours of extubation (if feasible). The following physiological and biological variables will be collected before and after the spontaneous breathing trial (SBT): mode of ventilation and settings, Arterial Blood Gas (ABG) results, heart rate, arterial blood pressure, peripheral capillary oxygen saturation (SpO2), respiratory rate, Glasgow Coma Score (GCS), temperature, fluid balance in the last 24 hours, Sequential Organ Failure Assessment (SOFA) score, and rapid shallow breathing index (RSBI). At the time of the ultrasound measurements, the following physiological variables will be collected: heart rate, arterial blood pressure, SpO2, respiratory rate, Glasgow Coma Score (GCS), cough, Intensive Care Delirium Screening Checklist (ICDSC), ambient air, oxygenation, use of non-invasive ventilation (NIV), level of dyspnea, level of comfort, nasal flaring, Medical Research Council (MRC) score, and the Respiratory Intensive Care Observation Scale (RICOS). Outcome data will be recorded including: extubation failure, use of NIV and/or high-flow nasal oxygen cannula post extubation, re-intubation, ICU discharge/re-admission status, and tracheostomy. A 7-day follow-up after ICU discharge will signify completion of the study.

ELIGIBILITY:
Inclusion Criteria:

* Invasive mechanical ventilation ≥ 48 hours
* Successful spontaneous breathing trial completed and extubation decided by the attending physician

Exclusion Criteria:

* Withholding or withdrawal of life support
* Patients under extracorporeal membrane oxygenation circuit
* Impossibility to perform ultrasound of the diaphragm of the two accessory muscles: neck surgery, C-spine collar, Halo vest, morbid obesity. Patients will be enrolled as long as access to at least two locations is feasible (intercostal, diaphragm, or sternocleidomastoid).
* Known (hemi) diaphragm paralysis

Min Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Extubated ICU patients.
Sampling Method: Non-Probability Sample
Enrollment: 124 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2018-03-31 (Actual); Study Completion 2018-03-31 (Actual)

PRIMARY OUTCOMES:
Comparison of the thickening fraction of each muscle (diaphragm, intercostal, and sternocleidomastoid) between 2 groups of patients regarding the occurrence of extubation failure risk and ICU readmission. | Up to 7 days after extubation

CONTACTS AND LOCATIONS:
Locations (1):
- St. Michael's Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Thille AW, Richard JC, Brochard L. The decision to extubate in the intensive care unit. Am J Respir Crit Care Med. 2013 Jun 15;187(12):1294-302. doi: 10.1164/rccm.201208-1523CI. PMID 23641924
- [Background] Matamis D, Soilemezi E, Tsagourias M, Akoumianaki E, Dimassi S, Boroli F, Richard JC, Brochard L. Sonographic evaluation of the diaphragm in critically ill patients. Technique and clinical applications. Intensive Care Med. 2013 May;39(5):801-10. doi: 10.1007/s00134-013-2823-1. Epub 2013 Jan 24. PMID 23344830
- [Background] Goligher EC, Laghi F, Detsky ME, Farias P, Murray A, Brace D, Brochard LJ, Bolz SS, Rubenfeld GD, Kavanagh BP, Ferguson ND. Measuring diaphragm thickness with ultrasound in mechanically ventilated patients: feasibility, reproducibility and validity. Intensive Care Med. 2015 Apr;41(4):642-9. doi: 10.1007/s00134-015-3687-3. Epub 2015 Feb 19. PMID 25693448
- [Background] Epstein SK, Ciubotaru RL, Wong JB. Effect of failed extubation on the outcome of mechanical ventilation. Chest. 1997 Jul;112(1):186-92. doi: 10.1378/chest.112.1.186. PMID 9228375
- [Background] Epstein SK, Ciubotaru RL. Independent effects of etiology of failure and time to reintubation on outcome for patients failing extubation. Am J Respir Crit Care Med. 1998 Aug;158(2):489-93. doi: 10.1164/ajrccm.158.2.9711045. PMID 9700126
- [Background] Parthasarathy S, Jubran A, Laghi F, Tobin MJ. Sternomastoid, rib cage, and expiratory muscle activity during weaning failure. J Appl Physiol (1985). 2007 Jul;103(1):140-7. doi: 10.1152/japplphysiol.00904.2006. Epub 2007 Mar 29. PMID 17395760
- [Background] DiNino E, Gartman EJ, Sethi JM, McCool FD. Diaphragm ultrasound as a predictor of successful extubation from mechanical ventilation. Thorax. 2014 May;69(5):423-7. doi: 10.1136/thoraxjnl-2013-204111. Epub 2013 Dec 23. PMID 24365607
- [Background] Ferrari G, De Filippi G, Elia F, Panero F, Volpicelli G, Apra F. Diaphragm ultrasound as a new index of discontinuation from mechanical ventilation. Crit Ultrasound J. 2014 Jun 7;6(1):8. doi: 10.1186/2036-7902-6-8. eCollection 2014. PMID 24949192
- [Background] Kim WY, Suh HJ, Hong SB, Koh Y, Lim CM. Diaphragm dysfunction assessed by ultrasonography: influence on weaning from mechanical ventilation. Crit Care Med. 2011 Dec;39(12):2627-30. doi: 10.1097/CCM.0b013e3182266408. PMID 21705883
- [Background] Jung B, Moury PH, Mahul M, de Jong A, Galia F, Prades A, Albaladejo P, Chanques G, Molinari N, Jaber S. Diaphragmatic dysfunction in patients with ICU-acquired weakness and its impact on extubation failure. Intensive Care Med. 2016 May;42(5):853-861. doi: 10.1007/s00134-015-4125-2. Epub 2015 Nov 16. PMID 26572511
- [Background] Adler D, Dupuis-Lozeron E, Richard JC, Janssens JP, Brochard L. Does inspiratory muscle dysfunction predict readmission after intensive care unit discharge? Am J Respir Crit Care Med. 2014 Aug 1;190(3):347-50. doi: 10.1164/rccm.201404-0655LE. No abstract available. PMID 25084264
- [Background] Goligher EC, Fan E, Herridge MS, Murray A, Vorona S, Brace D, Rittayamai N, Lanys A, Tomlinson G, Singh JM, Bolz SS, Rubenfeld GD, Kavanagh BP, Brochard LJ, Ferguson ND. Evolution of Diaphragm Thickness during Mechanical Ventilation. Impact of Inspiratory Effort. Am J Respir Crit Care Med. 2015 Nov 1;192(9):1080-8. doi: 10.1164/rccm.201503-0620OC. PMID 26167730
- [Background] Cala SJ, Kenyon CM, Lee A, Watkin K, Macklem PT, Rochester DF. Respiratory ultrasonography of human parasternal intercostal muscle in vivo. Ultrasound Med Biol. 1998 Mar;24(3):313-26. doi: 10.1016/s0301-5629(97)00271-8. PMID 9587987
- [Background] Jesus FM, Ferreira PH, Ferreira ML. Ultrasonographic measurement of neck muscle recruitment: a preliminary investigation. J Man Manip Ther. 2008;16(2):89-92. doi: 10.1179/106698108790818486. PMID 19119393
- [Background] Frutos-Vivar F, Ferguson ND, Esteban A, Epstein SK, Arabi Y, Apezteguia C, Gonzalez M, Hill NS, Nava S, D'Empaire G, Anzueto A. Risk factors for extubation failure in patients following a successful spontaneous breathing trial. Chest. 2006 Dec;130(6):1664-71. doi: 10.1378/chest.130.6.1664. PMID 17166980
- [Background] Thille AW, Harrois A, Schortgen F, Brun-Buisson C, Brochard L. Outcomes of extubation failure in medical intensive care unit patients. Crit Care Med. 2011 Dec;39(12):2612-8. doi: 10.1097/CCM.0b013e3182282a5a. PMID 21765357
- [Background] Thille AW, Cortes-Puch I, Esteban A. Weaning from the ventilator and extubation in ICU. Curr Opin Crit Care. 2013 Feb;19(1):57-64. doi: 10.1097/MCC.0b013e32835c5095. PMID 23235542